CLINICAL TRIAL: NCT03356171
Title: Combination of Cardiac Coherence to Physical Activity
Brief Title: Cardiac Coherence Combined With Personal Physical Activity in Patients With Cancer
Acronym: APACCHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017/CHU/06
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Physical Activity; Cancer; Hematologic Diseases
MeSH Terms: conditions — Motor Activity; Neoplasms; Hematologic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac Coherence (Experimental): Patients participate to Adapted physical activity sessions and to cardiac coherence sessions
  Interventions: Procedure: Cardiac Coherence
- Adapted Physical Activity (Active Comparator): Patients only participate to Adapted physical activity sessions
  Interventions: Procedure: Adapted Physical Activity

INTERVENTIONS:
Procedure: Cardiac Coherence — * 10 sessions of HRV-BF (45mn) weekly over 12 weeks. HRV-BF is a cognitive behavioural therapy consisting on stress management training based on breathing. We use the SYMBIOLINE PC software to record the heart rate variability biofeedback, with an infrared plethysmograph sensor. The sensor is put on the finger, and the patient's HRV pattern is displayed in real time.
  * 24 APA sessions (1.5h) bi-weekly over 12 weeks. Each session includes aerobic exercises (walk, step) and resistant exercises (muscular reinforcement). This program is built on previous cancer studies to make it effective.
  Arms: Cardiac Coherence
Procedure: Adapted Physical Activity — - 24 APA sessions (1.5h) bi-weekly over 12 weeks. Each session includes aerobic exercises (walk, step) and resistant exercises (muscular reinforcement). This program is built on previous cancer studies to make it effective.
  Arms: Adapted Physical Activity

SUMMARY:
APACCHE (Adapted Physical Activity and Cardiac Coherence in HEmatologic patients) study investigates effects of heart rate variability biofeedback training, combined with classical adapted physical activity, on health-related quality of life in patients previously treated for hematologic malignancies. It is a prospective, randomized clinical trial from University Hospital of Reunion Island. The main objective is evaluated with QLQ-C30 survey score differences.

DETAILED DESCRIPTION:
Hematologic malignancies are aggressive cancers with significant long-term effects on physical and psychological health, due to the disease itself or aggressive treatments. Physical activity, with specific treatments, improves physical and psychological health in solid tumors patients. However, in hematologic malignancies, there is unsatisfactory quality of evidence that physical activity alone improves the various dimensions of quality of life.

Recent studies on heart-brain connections suggest that a high level of coherence in the heart rate variability may induce psychophysiological positive effects. Cardiac coherence is reached when the heart rhythm pattern becomes sine-wave-like at a frequency around 0.1 Hz. This status can be increased by the mean of deep and slow breathing control and/or positive emotions. By using a heart rate variability biofeedback training, previous studies have shown effects on physiological variables such as reduction of blood pressure or increase of vagal heart rate control, and also on psychological variables such as reduction of stress, anxiety, and depression.

The APACCHE protocol investigate if cardiac coherence biofeedback training, associated with an adapted physical activity program, can improve health related quality of life in adult hematologic patients.

70 patients are randomly assigned to receive either ten sessions of cardiac coherence biofeedback (CC-BF) and the adapted physical activity program (APA) or just APA. Both interventions are conducted simultaneously over 12 weeks, with 10 sessions of CC-BF (45mn) weekly and 24 sessions of APA (1h30) bi-weekly.

Data are collected at enrollment(T1), at 6 weeks (T2), at intervention ending at 12 weeks (T3) and after a 24 weeks follow-up (T4).

ELIGIBILITY:
Inclusion Criteria:

* All patients, previously treated and in remission for an Hematologic malignancy, in whom APA is indicated.
* Adult patients aged 18-65 yo
* Followed at South University Hospital of La Réunion Island
* Previously treated for Hematologic Malignancy, and in Remission (complete or partial)
* 6 months or less since last treatment
* Hemoglobin steady ≥ 90g/L
* In whom APA is prescribed
* Ability to give oral informed consent
* French understanding

Exclusion Criteria:

* With contraindication for APA
* Under anti-arhythmic or beta-blocker drugs
* Cardiac insufficiency (Left ventriculi Ejection Fraction less than 40%)
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | on week 12
  Health-related quality is assessed by the Quality of Life Questionnaire dedicated to cancer patients and including 30 items (QLQ-C30) developed by the European Organization for Research and Treatment of Cancer (EORTC). This questionnaire is a multimodal construct, typically including physical, emotional and psychological health issues; evaluated with the QLQ-C30 survey of the European Organization for Research and Treatment of Cancer.
  QLQ-C30 items are coded with the same response categories as items 6 to 28, namely "Not at all", "A little", "Quite a bit" and "Very much." Score ranges from 0 to 100, with higher score indicating higher levels of quality of life.

SECONDARY OUTCOMES:
Fatigue improvement | through study completion: initially (T1), at 6 weeks (T2), 12 weeks (T3) and after at 24 weeks (T4) follow-up
  Fatigue improvement is assessed by multidimensional fatigue inventory (MFI-20 survey).
  MFI-20 consists of five subscales used to express: general fatigue, physical, reduced activities, reduced motivation, mental fatigue.
  Each scale contains four items for which the person had to indicate the extent the items describe their situations in the recent few days on a 5-point Likert scale, ranging from "yes, that is true" to "no, that is not true" Scores on each subscale range from 4 to 20, with higher scores indicating higher levels of fatigue.
Anxiety and depression improvement with Hospital Anxiety and Depression Scale (HADS) survey | through study completion: initially (T1), at 6 weeks (T2), 12 weeks (T3) and after at 24 weeks (T4) follow-up
  Anxiety and depression improvement is assessed by HADS survey. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3: a person can score between 0 and 21 for either anxiety or depression.
  Higher scores indicate higher levels of depression or anxiety
Cardiac coherence improvement | through study completion: initially (T1), at 6 weeks (T2), 12 weeks (T3) and after at 24 weeks (T4) follow-up
  Increased percentage of cardiac coherence is measured with SYMBIOLINE software

CONTACTS AND LOCATIONS:
Overall Officials: Quentin CABRERA, MD, Principal Investigator — Centre Hospitalier Universitaire de La REUNION, France
Locations (1):
- Centre Hospitalier Universitaire de La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fournie C, Bouscaren N, Dalleau G, Lenclume V, Mohr C, Zunic P, Cabrera Q, Verkindt C. Adapted physical activity and cardiac coherence in hematologic patients (APACCHE): study protocol for a randomized controlled trial. BMC Sports Sci Med Rehabil. 2020 Mar 14;12:18. doi: 10.1186/s13102-020-00170-3. eCollection 2020. PMID 32190333